CLINICAL TRIAL: NCT06136793
Title: HomeStyles: Shaping HOME Environments and LifeSTYLE Practices to Reduce Cardiometabolic Disease Risk in Adults of Chinese Heritage Living in the United States
Brief Title: HomeStyles-Adults of Chinese Heritage
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Carol Byrd-Bredbenner, PhD, RD, FAND, Distinguished Professor of Nutrition, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro2020001192a; P50MD017356 (NIH)
Record Dates: First submitted 2023-11-08; First posted 2023-11-18 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Healthy Lifestyle; Home Environment Related Disease; Cardiometabolic Disease; Systemic Inflammatory Response; Health Behavior; Dietary Habits; Physical Inactivity; Self Efficacy; Gut Microbiota; Diabetes Mellitus
Keywords: Chinese heritage; Asian; Cardiometabolic disease; China; Chinese; Chronic disease; Health behavior; Dietary intake; physical activity; home environment; inflammation; randomized control trial; body mass index; hypertension; diabetes mellitus; health disparities; family; sleep; self efficacy
MeSH Terms: conditions — Health Behavior; Feeding Behavior; Sedentary Behavior; Diabetes Mellitus; Chronic Disease; Motor Activity; Inflammation; Hypertension

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Participant
Masking Description: concurrent treatments different in subject matter but equal in nonspecific treatment effects
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Healthy HomeStyles (Experimental): Online educational intervention
  Interventions: Behavioral: HomeStyles-China
- Active Comparator: Safe HomeStyles (Active Comparator): Online educational intervention
  Interventions: Behavioral: HomeStyles-China

INTERVENTIONS:
Behavioral: HomeStyles-China — 2-arm ~10 week educational intervention

SUMMARY:
Individuals of Chinese heritage are the largest and fastest growing segment of the US Asian population. US Chinese have sociodemographic characteristics and culture that differ substantially from other US Asians, and therefore, differ in social determinants of health, health status, and disease risk. US Chinese adults are at increased risk for cardiometabolic disease, related conditions (obesity, type 2 diabetes mellitus, hypertension), and systemic inflammation that promotes disease onset and progression. Immigration to a new country can substantially impact the gut microbiome which may promote systemic inflammation. Pilot interventions indicate a high-fiber diet rich in whole grains reduced inflammation and improved obesity. Additionally, the United States Department of Agriculture (USDA) supported, evidence-based HomeStyles intervention has demonstrated feasibility, acceptability, and efficacy in improving lifestyle behaviors and home environments associated with obesity risk in families. A lack of linguistically, culturally tailored interventions to their specific health needs makes it difficult for US Chinese to implement healthy lifestyle behaviors and reduce health risks. Interventions tailored for US Chinese that could attenuate modifiable cardiometabolic risk factors, understand physiological sequelae, and bridge health equity are not currently available. Thus, the overall goal of this project is to test the efficacy of HomeStyles in improving health outcomes in US Chinese. Project aims are to: A) Culturally adapt the HomeStyles intervention through community-engaged approaches. B) Conduct a 10-week, 2-armed Randomized Controlled Trial (RCT) to test HomeStyles intervention efficacy on health outcomes (dietary intake, physical activity, self-efficacy, HbA1C, waist circumference, and BMI), hypothesizing that participants randomized to the treatment condition will have greater improvements in health outcomes than control comparators. C) Examine associations between intervention participation and gut microbiota/systemic inflammation and test hypotheses that a whole-grain rich diet adopted by those in the intervention group will increase anti-inflammatory gut bacteria, reduce inflammatory gut bacteria, and lower systemic inflammation.

DETAILED DESCRIPTION:
The aim of the HomeStyles-China RCT is to determine whether this novel, culturally tailored intervention enables and motivates adults of Chinese heritage living in the United States to shape their home environments and weight-related lifestyle practices (i.e., diet, exercise, sleep) to reduce risk for cardiometabolic disease, related conditions, and systemic inflammation more than those in the control condition. RCT Design CONSORT guidelines extension for social and psychological intervention trials will be used to generate a participant flow diagram and report RCT enrollment and retention data. Interested participants will begin by completing a short eligibility screener survey. Eligible participants who give informed consent will have immediate access to the baseline survey. Those who complete the baseline survey, meet survey plausibility checks, and complete the registration page (e.g., provide name and contact information) will be enrolled in the RCT. Enrolled participants will be systematically randomized by computer by alternating assignment to the experimental or attention control study condition. Recruitment materials and the bona fide treatment to be delivered to the attention control group are designed to blind participant assignment to study condition. Participants will receive intervention materials starting immediately after registration and at weekly intervals for 9 weeks. In week 10 of the study, participants will be invited to take the post survey to assess intervention effects. Approximately 12 weeks after participants complete the post survey, they will be invited to take the follow-up survey to assess longer-term intervention effects. Participants who complete the baseline survey will be invited to provide blood and/or fecal samples; those who consent will have the opportunity to provide samples coincident with the post and follow-up surveys. If the participant does not have a cardiometabolic condition but indicates another adult living in the household has a condition, the other adult also will be recruited to provide blood and/or fecal samples.

Each week of the 9-week intervention, participants will be encouraged to spend about 15 minutes reviewing intervention materials; think about the changes like those suggested in the materials that could help their families; and implement 1 or 2 easy, quick, low-cost changes in their homes. Intervention materials (described in a subsequent section) provided each week for 9 weeks include an electronic informational guide for participants, tracker to list guide-related goals for the week and monitor progress toward them, and 3 to 4 encouraging nudges delivered by text and email.

Participant progress through the RCT will be monitored by project staff by observing their visits to the website. Bilingual staff will be trained in customer service strategies and instructed to quickly address any participant queries using scripted responses to ensure equitable care across study groups. Participants will receive modest stipends that increase in value after they complete each survey. Those consenting to blood and/or fecal analyses also will receive modest stipends increasing in value from baseline, to post, to follow-up.

HomeStyles-China is an intervention program that enables and motivates adults to shape their lifestyle behavioral practices and home environments to create and support optimal health and reduce risk factors for and markers of obesity and related chronic conditions. HomeStyles is designed for adults to implement within their homes in partnership with other family members. The home environment is targeted because it plays a dominant role in families, especially those with children and teens who are developing eating and physical activity patterns and these patterns track across the growing years into adulthood. Adults are the family household food gatekeepers and create the structure/lifestyle environment within the home, and thus, strongly influence health protective behaviors of other family members. In addition, adults need more opportunities to gain relevant, practical, non-judgmental obesity prevention information that is easily implemented in their homes and hectic lifestyles.

Experimental Group Intervention: The HomeStyles experimental group intervention materials (i.e., "Healthy" HomeStyles-China) were designed to be congruent with White House and Institute of Medicine (IOM) recommendations for home-centered obesity prevention interventions and critical elements for effective interventions (e.g., interventions are positive, culturally sensitive, supportive of family interactions; develop realistic, effective plans that empower families). Like HomeStyles for preschoolers and HomeStyles-2 for middle childhood intervention materials, HomeStyles-China experimental group intervention materials provide intensive, interactive, fun, non-judgmental opportunities for adults to shape their home environments and lifestyle practices to protect family health. They also promote positive strategies and changes that adults can control in their environments to reduce risk for cardiometabolic disease and related conditions. A positive approach teaches individuals what they can do (eat more fruits) rather than giving prohibitions (cut out fries). Substantial evidence supports preference for positive messages and the value of promoting positive vs restrictive behaviors to achieve health goals.

Intervention Content. Key factors contributing to cardiometabolic disease risk that can be suitably addressed in the home environment identified for inclusion in the intervention materials are inadequate intake of fruits and vegetables, infrequent family meals, excessive consumption of sugar-sweetened beverages, large portion sizes, irregular breakfast consumption, inadequate intake of whole grain foods, limited physical activity, and inadequate sleep.

Attention Control Intervention The attention control intervention will use bona fide, credible materials that are structurally equivalent to the experimental group. The attention control treatment will be credible in that it focuses on a topic fitting the description of the study recruitment materials (i.e., shaping homes and lifestyles to help families be even happier and healthier) yet providing distinctly different, non-overlapping content (i.e., home safety) devoid of the RCT "active" ingredient (i.e., content related to cardiometabolic disease reduction). The attention control intervention materials include the same components as those used in the experimental group (i.e., instructional guides, trackers, nudges) with the content focused on home safety.

The Safe HomeStyles guides focus on indoor air quality, mold & moisture, hazardous household products, carbon monoxide, home safety, foodborne illness, lead safety, and safe food storage. The Safe HomeStyles materials have an appearance and structure similar to those in the experimental group.

Instruments The study survey, "Home Obesogenicity Measures of EnvironmentS"-Families of Chinese Heritage (HOMES-China), will be used to collect baseline, post, and follow-up data in the RCT. The Social Cognitive Theory along with the key concepts addressed in the HomeStyles-China guides provided the framework for identification of cognitions, behaviors, and aspects of the home environment to be assessed. Online survey collection procedures will be used to collect baseline, post, and follow-up self-report data. The survey will collect sociodemographic characteristics, health status; cardiometabolic health-related cognitions and behaviors; and cardiometabolic health-related characteristics of the home environment. When the participant does not have a cardiometabolic condition but another adult in the family does, sociodemographic characteristics, health status, and cardiometabolic-related health behaviors of the other adult will be collected. A subset of participants (and when applicable, another adult family member) will be invited to provide a blood sample and fecal sample.

ELIGIBILITY:
Inclusion Criteria:

* adult of Chinese heritage >30 years with a self-reported cardiometabolic condition or living with an adult (spouse/partner, parent) with a cardiometabolic condition; primary food gatekeeper in the household (i.e., makes all or most decisions related to family food choices); has regular Internet access, read English and/or Chinese, and resides in New York/New Jersey metro area

Exclusion Criteria:

* Does not fit inclusion criteria

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Participant Health-related behaviors: Fruit/Vegetable/Fiber Intake (servings/day) | Pre-intervention (baseline), post-intervention (~10 weeks after baseline), follow-up (~12 weeks after post-intervention)
  Dietary intake: Block Fruit/Vegetable/Fiber Screener servings/day; possible range 0 to infinity
Participant Health-related behaviors: Sugar-sweetened Beverage Intake (servings/day) | Pre-intervention (baseline), post-intervention (~10 weeks after baseline), follow-up (~12 weeks after post-intervention)
  Dietary intake: HOMES Sugar-sweetened beverage Intake servings/day; possible range 0 to infinity
Participant Health-related behaviors: Physical Activity Level | Pre-intervention (baseline), post-intervention (~10 weeks after baseline), follow-up (~12 weeks after post-intervention)
  Physical activity: Streamlined International Physical Activity Questionnaire; possible range 0 to 49; 49 is highest
Participant Health-related behaviors: Self-Efficacy for Health Behaviors | Pre-intervention (baseline), post-intervention (~10 weeks after baseline), follow-up (~12 weeks after post-intervention)
  HOMES Self-Efficacy for Engaging in Healthy Cardiometabolic Behaviors; possible score range 1 to 5; 5 is highest
Participant Cardiometabolic Disease Markers: Diabetes Risk | Pre-intervention (baseline), post-intervention (~10 weeks after baseline), follow-up (~12 weeks after post-intervention)
  HbA1c; percentage; normal below 5.7%; prediabetes 5.7 to 6.4%; diabetes 6.5% or above
Participant Cardiometabolic Disease Markers: Height (for BMI calculation) | Pre-intervention (baseline), post-intervention (~10 weeks after baseline), follow-up (~12 weeks after post-intervention)
  Height (in cm)
Participant Cardiometabolic Disease Markers: Weight (for BMI calculation) | Pre-intervention (baseline), post-intervention (~10 weeks after baseline), follow-up (~12 weeks after post-intervention)
  Weight (in kg)
Participant Cardiometabolic Disease Markers: Waist circumference | Pre-intervention (baseline), post-intervention (~10 weeks after baseline), follow-up (~12 weeks after post-intervention)
  Waist circumference (in cm) for central adiposity assessment

SECONDARY OUTCOMES:
Participant Health-related Behavior: Sleep duration | Pre-intervention (baseline), post-intervention (~10 weeks after baseline), follow-up (~12 weeks after post-intervention)
  Participant sleep duration: Pittsburgh Sleep Quality Index; Sleep Duration Component; possible score 0 to 24 hours
Participant Cardiometabolic Disease Marker: Lipid | Pre-intervention (baseline), post-intervention (~10 weeks after baseline), follow-up (~12 weeks after post-intervention)
  Lipid panel: total cholesterol, triglycerides, HDL, LDL
Participant Cardiometabolic Disease Marker: Inflammation | Pre-intervention (baseline), post-intervention (~10 weeks after baseline), follow-up (~12 weeks after post-intervention)
  hsCRP
Other adult living in household with a cardiometabolic condition, if participant does not have cardiometabolic condition: Fruit/Vegetable/Fiber Intake (servings/day) | Pre-intervention (baseline), post-intervention (~10 weeks after baseline), follow-up (~12 weeks after post-intervention)
  Dietary intake: Block Fruit/Vegetable/Fiber Screener servings/day; possible range 0 to infinity
Other adult living in household with a cardiometabolic condition, if participant does not have cardiometabolic condition: Sugar-Sweetened Beverage Intake (servings/day) | Pre-intervention (baseline), post-intervention (~10 weeks after baseline), follow-up (~12 weeks after post-intervention)
  Dietary intake: HOMES Sugar-sweetened beverage Intake servings/day; possible range 0 to infinity
Other adult living in household with a cardiometabolic condition, if participant does not have cardiometabolic condition: Physical Activity Level | Pre-intervention (baseline), post-intervention (~10 weeks after baseline), follow-up (~12 weeks after post-intervention)
  Physical activity: Streamlined International Physical Activity Questionnaire; possible range 0 to 49; 49 highest
Other adult living in household with a cardiometabolic condition, if participant does not have cardiometabolic condition: Sleep Duration Behaviors | Pre-intervention (baseline), post-intervention (~10 weeks after baseline), follow-up (~12 weeks after post-intervention)
  Other adult sleep duration: Pittsburgh Sleep Quality Index; Sleep Duration Component; possible score 0 to 24 hours
Other adult living in household with a cardiometabolic condition, if participant does not have cardiometabolic condition Cardiometabolic Disease Markers: Lipid | Pre-intervention (baseline), post-intervention (~10 weeks after baseline), follow-up (~12 weeks after post-intervention)
  Lipid panel: total cholesterol, triglycerides, HDL, LDL
Other adult living in household with a cardiometabolic condition, if participant does not have cardiometabolic condition Cardiometabolic Disease Markers: Inflammation | Pre-intervention (baseline), post-intervention (~10 weeks after baseline), follow-up (~12 weeks after post-intervention)
  hsCRP
Other adult living in household with a cardiometabolic condition, if participant does not have cardiometabolic condition Diabetes Risk | Pre-intervention (baseline), post-intervention (~10 weeks after baseline), follow-up (~12 weeks after post-intervention)
  HbA1c; percentage; normal below 5.7%; prediabetes 5.7 to 6.4%; diabetes 6.5% or above
Other adult living in household with a cardiometabolic condition, if participant does not have cardiometabolic condition: Height | Pre-intervention (baseline), post-intervention (~10 weeks after baseline), follow-up (~12 weeks after post-intervention)
  Height (in cm) for BMI calculation
Other adult living in household with a cardiometabolic condition, if participant does not have cardiometabolic condition: Weight | Pre-intervention (baseline), post-intervention (~10 weeks after baseline), follow-up (~12 weeks after post-intervention)
  Weight (in kg) for BMI Calculation
Other adult living in household with a cardiometabolic condition, if participant does not have cardiometabolic condition: Waist Circumference | Pre-intervention (baseline), post-intervention (~10 weeks after baseline), follow-up (~12 weeks after post-intervention)
  Waist circumference (in cm) for central adiposity assessment
Household Supports for cardiometabolic disease reduction measures: Environmental Supports | Pre-intervention (baseline), post-intervention (~10 weeks after baseline), follow-up (~12 weeks after post-intervention)
  HOMES Environment Supports for Cardiometabolic Health; possible score 1 to 5; 5 highest
Household Supports for cardiometabolic disease reduction measures: Family Collective-Efficacy | Pre-intervention (baseline), post-intervention (~10 weeks after baseline), follow-up (~12 weeks after post-intervention)
  HOMES Family Collective-Efficacy; possible score 1 to 5; 5 highest

CONTACTS AND LOCATIONS:
Overall Officials: Carol Byrd-Bredbenner, Principal Investigator — Rutgers University

IPD SHARING:
Plan to Share IPD: Yes
Deidentified primary and secondary outcome data will be shared after study data are published and upon request
Supporting Information: Study Protocol
Time Frame: At the conclusion of the study after study data are published
Access Criteria: Request for data access to PI